CLINICAL TRIAL: NCT02794168
Title: Efficacy of VAS203 (Ronopterin) in Patients With Moderate and Severe Traumatic Brain Injury - (NOSTRA Phase III Trial): A Confirmatory, Placebo-controlled, Randomised, Double Blind, Multi-centre Study
Brief Title: Efficacy of VAS203 (Ronopterin) in Patients With Moderate and Severe Traumatic Brain Injury
Acronym: NOSTRA-III
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: veriNOS operations GmbH (Industry)
Collaborators: ICON plc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: VAS203/III/1/04
Record Dates: First submitted 2016-05-31; First posted 2016-06-08 (Estimated); Last update posted 2021-10-11 (Actual); Status verified 2021-10

CONDITIONS: Traumatic Brain Injury
MeSH Terms: conditions — Brain Injuries, Traumatic | interventions — 4-amino-tetrahydrobiopterin; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- VAS203 (Ronopterin) (Experimental): Intravenous infusion of 17 mg/kg VAS203 over 48 hours, daily dose 8.5 mg/kg
  Interventions: Drug: VAS203
- Saline (Placebo Comparator): Intravenous infusion of physiological saline over 48 hours
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: VAS203 — Treatment
  Other Names: Ronopterin
  Arms: VAS203 (Ronopterin)
Drug: Saline — Placebo
  Arms: Saline

SUMMARY:
This study evaluates the efficacy of an infusion of Ronopterin (VAS203) on clinical outcome in patients with moderate and severe traumatic brain injury. Half of the participants will receive Ronopterin (VAS203), while the other half will receive placebo.

DETAILED DESCRIPTION:
Severe and moderate traumatic brain injury (TBI) constitutes a major health problem. TBI is the leading cause of death and disability among young adults in developed countries, and the incidence in the elderly population is increasing.

Neurological damage after TBI is caused not only by the accident itself, but evolves afterwards. The posttraumatic secondary injury includes - among others - inflammation and oedema formation with subsequent increase of intracranial pressure. A key molecule in these processes is the gas nitric oxide, which is produced in excess during neuroinflammation.

Ronopterin (VAS203) is an inhibitor of nitric oxide synthase. Ronopterin reduces excess nitric oxide production and subsequent secondary injury.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent from patient's legal guardian or legal representative or deferred consent procedure, according to local requirements
2. 18 - 60 years of age, inclusive
3. Expected to survive more than 24 hours after admission
4. Traumatic Brain Injury (TBI) within the last 18 hours (infusion must not start earlier than 6 hours after the injury)
5. TBI with Glasgow Coma Score (GCS) ≥ 3 requiring intracranial pressure (ICP) monitoring according to the assessment of the treating physician.
6. Catheter placement (intraventricular or intraparenchymal, only) for monitoring and management of increased ICP
7. Systolic blood pressure ≥ 100 mmHg
8. Females of child-bearing potential must have a negative pregnancy test

Exclusion Criteria:

1. Penetrating head injury (e.g. missile, stab wound)
2. Concurrent, but not pre-existing, spinal cord injury
3. Bilateral fixed and dilated pupil (> 4 mm)
4. Cardiopulmonary resuscitation performed post injury, or extracranial injuries causing continuing bleeding likely to require multiple transfusions (> 4 units red blood cells)
5. Coma due to an exclusive epidural hematoma (lucid interval and absence of structural brain damage on CT scan)
6. Coma suspected to be primarily due to other causes than head injury (e.g. drug overdose intoxication, drowning/near drowning)
7. Known or CT scan evidence of pre-existing major cerebral damage
8. Patients who cannot be monitored with regard to their recovery (eGOS-I and QOLIBRI)
9. Patients and relatives of patients who don´t understand/speak Spanish, or English, or French, or German
10. Decompressive craniectomy, planned prior to randomisation
11. Polytraumatic patients with Injury Severity Score non-head > 18
12. Rhabdomyolysis with Creatine Kinase > 5000 IU/L
13. Injuries to ascending aorta and/or carotid arteries and vertebral arteries
14. Serum creatinine values > 1.2 mg/dL (106 µmol/L) (women), or > 1.5 mg/dL (133 µmol/L) (men)
15. Estimated glomerular filtration rate (eGFR) < 60 mL/min as calculated by Chronic Kidney Disease Epidemiology Collaboration Formula
16. BMI < 18.5 kg/m2 and > 40 kg/m2, Body weight > 110 kg
17. Any severe concomitant condition (cancer; hematologic, renal, hepatic, coronary disease; major psychiatric disorder; alcohol or drug abuse), that can be ascertained at admission
18. Known to have received an experimental drug within 4 weeks prior to current injury

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 224 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
extended Glasgow Outcome Scale | 6 months
  clinical outcome questionnaire

SECONDARY OUTCOMES:
Quality of life after brain injury (QOLIBRI) | 6 months
  clinical outcome questionnaire
QOLIBRI overall scale | 6 months
  clinical outcome questionnaire
extended Glasgow Outcome Scale | 3 months
  clinical outcome questionnaire
QOLIBRI overall scale | 3 months
  clinical outcome questionnaire
Therapy Intensity Level | 14 days
  Daily recording of score for therapeutic measures
Number of decompressive craniectomies | 14 days
  Number of decompressive craniotomies on both hemispheres

OTHER OUTCOMES:
Adverse Events | 14 days
  Number of adverse events related to treatment
Renal function | 14 days
  Number of patients exhibiting acute kidney injury according Acute Kidney Injury Network criteria
Mortality | 6 Months
  Mortality 6 months after traumatic brain injury

CONTACTS AND LOCATIONS:
Overall Officials: Erich Schmutzhard, Prof. MD, Principal Investigator — Medical University Innsbruck
Locations (29):
- Austria (3):
  - Universitätsklinik für Neurochirurgie, Graz
  - Neurologie und Neurochirurgie Medizinische Universität Innsbruck, Innsbruck
  - Klinik für Allgemeine Anästhesie und Intensivmedizin AKH Wien, Vienna
- France (4):
  - Hôpital Pellegrin Service de réanimation traumatologique et chirurgicale, Bordeaux
  - Hopital Gabriel Montpied, Clermont-Ferrand
  - Pôle Anesthésie Réanimation Douleur Urgence, Nîmes
  - HIA Sainte-Anne Boulevard Sainte-Anne, Toulon
- Germany (14):
  - Charite Virchow-Klinikum, Berlin
  - Berufsgenossenschaftliche Kliniken Bergmannsheil Klinik für Neurochirurgie, Bochum
  - Allgemeines Krankenhaus Celle Neurotraumatologie, Celle
  - Universitätsklinikum Düsseldorf Neurochirurgische Klinik, Düsseldorf
  - Klinik für Neurochirurgie Universität Frankfurt, Frankfurt
  - Universitätsklinikum Göttingen Klinik für Neurochirurgie, Göttingen
  - Berufsgenossenschaftliche Kliniken Bergmannstrost Halle Klinik für Neurochirurgie, Halle
  - Universitätsklinikum Hamburg-Eppendorf Klinik und Poliklinik für Neurochirurgie, Hamburg
  - Medizinische Hochschule Hannover Klinik für Neurochirurgie, Hanover
  - Neurochirurgische Universitätsklinik Heidelberg, Heidelberg
  - Universitätsklinikum des Saarlands, Homburg
  - Universitätsklinikum Jena Klinik und Poliklinik für Neurochirurgie, Jena
  - Universitätsklinikum Schleswig-Holstein Klinik für Neurochirurgie, Kiel
  - Universitätsklinikum Leipzig Klinik und Poliklinik für Neurochirurgie, Leipzig
- Spain (4):
  - Vall d'Hebron University Hospital Department of Neurosurgery, Barcelona
  - Hospital General Universitario, Elche
  - Hospital 12 de Octubre, Madrid
  - Son Espases University Hospital, Palma
- United Kingdom (4):
  - Queen Elizabeth Hospital Birmingham, Birmingham
  - NHS Lothian University of Edinburgh, Edinburgh
  - Kings College Hospital London, London
  - Southampton University Hospital Division of Clinical Neurosciences, Southampton

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Stover JF, Belli A, Boret H, Bulters D, Sahuquillo J, Schmutzhard E, Zavala E, Ungerstedt U, Schinzel R, Tegtmeier F; NOSTRA Investigators. Nitric oxide synthase inhibition with the antipterin VAS203 improves outcome in moderate and severe traumatic brain injury: a placebo-controlled randomized Phase IIa trial (NOSTRA). J Neurotrauma. 2014 Oct 1;31(19):1599-606. doi: 10.1089/neu.2014.3344. Epub 2014 Jul 28. PMID 24831445
- [Derived] Tegtmeier F, Schinzel R, Beer R, Bulters D, LeFrant JY, Sahuquillo J, Unterberg A, Andrews P, Belli A, Ibanez J, Lagares A, Mokry M, Willschke H, Fluh C, Schmutzhard E; NOSTRA Investigators. Efficacy of Ronopterin (VAS203) in Patients with Moderate and Severe Traumatic Brain Injury (NOSTRA phase III trial): study protocol of a confirmatory, placebo-controlled, randomised, double blind, multi-centre study. Trials. 2020 Jan 14;21(1):80. doi: 10.1186/s13063-019-3965-4. PMID 31937347